CLINICAL TRIAL: NCT02876666
Title: Spinal Cord Injury Virtual Coach to Promote Self-Care in Pressure Ulcer Prevention
Brief Title: Spinal Cord Injury Virtual Coach RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-33729; 324644 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Health Behavior
MeSH Terms: conditions — Spinal Cord Injuries; Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coach Intervention (Experimental)
  Interventions: Behavioral: SCI Virtual Coach
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: SCI Virtual Coach — Participants are given a computer with the SCI Virtual Coach program and are asked to interact with the Coach daily for 2 months.
  Arms: Coach Intervention

SUMMARY:
The SCI Virtual Coach study has developed an on-screen, human-like character that will provide support, education and coaching to adults with spinal cord injury (SCI) to aid in the prevention of serious secondary conditions like pressure ulcers. In a randomized controlled trial, participants assigned to "the Coach" intervention will have a touch-screen computer placed in their homes and be asked to interact with the Coach on a daily basis for 2 months. Participants will be asked to complete surveys at baseline and 2 months.

The SCI Virtual Coach study aims to measure how accessible and usable participants feel the Coach is, as well as participants' adherence to the Coach's instructions. It will also gauge how effective the Coach is in changing self-care knowledge, health care behaviors, self-efficacy for self-care, and perception of social support in participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of physician-confirmed chronic spinal cord injury diagnosis
* Injured within the last 6 months -10 years
* Speaks and understands conversational English
* Lives within approximately 1 hour of Boston, MA

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Expected to live less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Standardized Usability Questionnaire | Report at 2 month exit survey
  Evaluates the participant's self-reported experiences with the Coach on a number of characteristics, including ease of use, repetitiveness, and overall satisfaction.

SECONDARY OUTCOMES:
Health Education Impact Questionnaire - Skill Technique Acquisition | Baseline and 2 months
  Self-report measure of the participant's feelings about their ability to do skin behavior tasks
Skin Care Behavior Compliance | Baseline and two months
  Self-report measure of compliance with behaviors to prevent skin care problems that lead to pressure ulcers

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Latham, PT, PhD, Principal Investigator — Boston University
Locations (1):
- New England Regional SCI Center, Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No